CLINICAL TRIAL: NCT02920086
Title: Improving Partnerships With Family Members of ICU Patients: The IMPACT Trial
Brief Title: Improving Partnerships With Family Members of ICU Patients
Acronym: IMPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Griffith University (Other)
Responsible Party: Principal Investigator, Daren K. Heyland, Principal Investigator, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IMPACT
Record Dates: First submitted 2016-09-19; First posted 2016-09-30 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Optics and Photonics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutrition Education Program (Experimental): Nutrition education for family members of an elderly critically ill patient
  Interventions: Behavioral: Nutrition Education Program
- Decision Support Program (Experimental): Decision support education for family members of an elderly critically ill patient
  Interventions: Other: Decision Support Program
- Usual Care (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Nutrition Education Program — * The OPTimal nutrition by Informing and Capacitating family members of best practices (OPTICS) intervention
  * Nutritional education will be provided to ICU patents' families by a dietitian
  * Tracking of nutritional information by family
  * Encouragement for families to advocate for two or more Oral Nutritional Supplements per day for the patients (approximately 400 kcal/day)
  Other Names: OPTICS
  Arms: Nutrition Education Program
Other: Decision Support Program — * Families will be provided with a web-based decision support tool (My ICU Guide)
  * Families will meet with the ICU medical team early in ICU stay to review goals of care
  Other Names: The REALISTIC-80 Decision Support Intervention; My ICU Guide
  Arms: Decision Support Program

SUMMARY:
The purpose of this study is to improve the outcomes of critically ill older patients and the health outcomes of their families by capacitating and partnering with families in optimizing patient/family centered care.

DETAILED DESCRIPTION:
There is a pressing need to improve the care of critically ill older patients. For critically ill patients who are frequently unable to participate in their own care and decision-making, partnering with their family members is particularly important for improving experiences and outcomes of care for both patients and families. However, the optimal means by which families engage in the role they play, and how best to capacitate them as advocates and partners in care while helping them maintain their own wellbeing, is not known.

The IMPACT trial will evaluate two interventions, each with a separate context, but similar in that they empower and support families; one focused on involvement in care, and the other focused on involvement in decision-making. The first is a nutrition intervention The OPTimal nutrition by Informing and Capacitating family members of best practices (OPTICs) intervention, a multi-faceted strategy to engage and empower family members to advocate for and audit best nutrition practices in their family members. The second is a decision support intervention. The REALISTIC-80 Decision Support Intervention, is a web-based tool (www.myicuguide.com) to support families in shared decision-making about goals of medical treatments.

The investigators propose to conduct a mixed methods multi-centre, open-label, randomized, clinical trial involving 3 groups (2 active interventions and a usual care group). The overall goal of this study is to demonstrate that the multi-faceted nutritional strategies that engage families in care of their family member tested in this trial will increase nutritional intake and optimize physical recovery in older critically ill patients at high nutrition risk.

ELIGIBILITY:
Inclusion Criteria for Patients:

1a) > 60 years of age OR

1b) 55 years to 59 years old with one or more of the following diagnoses:

* Chronic obstructive lung disease - 2 of the 4 of: baseline PaCO2 of > 45 torr, cor pulmonale; respiratory failure episode within the preceding year; forced expiratory volume in 1 sec <0.5 L.
* Congestive heart failure - New York Heart Association class IV symptoms and left ventricular ejection fraction < 25%.
* Cirrhosis - confirmed by imaging studies or documentation of esophageal varices and one of three conditions: a) hepatic coma, b) Child's class C liver disease, or c) Child's class B liver disease with gastrointestinal bleeding.
* Cancer - metastatic cancer or stage IV lymphoma.
* End-stage dementia (inability to perform all ADLs, mutism or minimal verbal output secondary to dementia, bed-bound state prior to acute illness) 2) Have a projected duration of ICU dependency of >72 hours from time of final assessment. We define ICU dependency as the need for one or more of the following:
* Mechanical ventilation
* Non-invasive ventilation
* Renal replacement therapy
* Vasopressors or
* Artificial nutrition because of their underlying illness

Exclusion Criteria for Patients:

* Patients who are not expected to remain alive in ICU for 72 hours after initial screening (physician judgment) or for whom life-sustaining treatments are expected to be withdrawn in the subsequent 72 hours (as sufficient time will be required for implementation of the study interventions)
* Uncomplicated elective surgical patients (regardless of age)
* Patients who have received organ transplantation during this hospitalization

Inclusion Criteria for Family Member:

* 18 years of age or older,
* present and expected to visit regularly (minimum about 3 times a week) while the patient is in hospital
* the nominated or legally appointed substitute decision-maker
* able to communicate in English (verbally and in writing).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-05-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional adequacy during the ICU stay | Up to 30 days in ICU
Consumption of Oral Nutritional Supplements | First four weeks once on ward
Intake on hospital wards (3 day calorie count) | First four weeks once on ward
Hand grip strength | At or before hospital discharge or up to 90 days
  Hydraulic hand dynamometer
Use of shared-decision making (OPTION tool) | Within first week in ICU
Change in decisional conflict | 1 week
  10-item Decisional Conflict Scale
Family satisfaction with decision-making | 1 week
Overall family satisfaction with ICU | At ICU discharge, an average of 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Daren Heyland, MD, Principal Investigator — Clinical Evaluation Research Unit
Locations (10):
- United States (5):
  - Phoenix VA Medical Center, Phoenix, Arizona
  - Barnes Jewish Hospital/Washington University, St Louis, Missouri
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Gold Coast Health, Gold Coast, Queensland, Australia
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Ottawa, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marshall AP, Van Scoy LJ, Chaboyer W, Chew M, Davidson J, Day AG, Martinez A, Patel J, Roberts S, Skrobik Y, Taylor B, Tobiano G, Heyland DK. A randomised controlled trial of a nutrition and a decision support intervention to enable partnerships with families of critically ill patients. J Clin Nurs. 2023 Sep;32(17-18):6723-6742. doi: 10.1111/jocn.16752. Epub 2023 May 9. PMID 37161555
- [Derived] Heyland DK, Davidson J, Skrobik Y, des Ordons AR, Van Scoy LJ, Day AG, Vandall-Walker V, Marshall AP. Improving partnerships with family members of ICU patients: study protocol for a randomized controlled trial. Trials. 2018 Jan 4;19(1):3. doi: 10.1186/s13063-017-2379-4. PMID 29301555